CLINICAL TRIAL: NCT02237352
Title: Physiopathogenic Mechanisms Involved in Diabetic Nephropathy, Looking for Prevention and Treatment Solutions
Brief Title: Mechanisms of Diabetic Nephropathy in Ecuador
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad Estatal de Milagro (Other)
Collaborators: Secretaría de Ciencia, Tecnología e Innovación (Senescyt) (Unknown); PROMETEO (Unknown)
Responsible Party: Sponsor
Other Study IDs: DN-HLV0178-DV
Record Dates: First submitted 2014-08-20; First posted 2014-09-11 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Nephropathy; Diabetes Mellitus; Kidney Diseases; Diabetic Kidney Disease; Chronic Kidney Disease
Keywords: Diabetes mellitus; Diabetic nephropathy; Social Factors; Biological Factors; VEGF-A; Tenascin C; Disease characterization; Mechanisms; Kidney; Chronic kidney disease; Secondary nephropathy; South America; Hispanics; Ecuador; Biomarkers
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Plasma and urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Subjects without diabetic nephropathy
- Diabetic nephropathy: Subjects with diabetic nephropathy

SUMMARY:
The prevalence of diabetes mellitus (DM) is increasing worldwide, suggesting that 45% of diabetics are undiagnosed. DM induces a kidney disease called diabetic nephropathy (DN) which is the largest single cause of end-stage renal disease and dialysis requirement. In South America the prevalence of DM and chronic kidney disease has increased, and great disparity exists among countries in regards to access to the dialysis treatment. It has been considerate that Hispanic origin increases the risk for DM. The South Americans have distinctive habits, culture, environment, behavior and genetic background and the factors involved in DN have not been defined yet. The early kidney lesions such as neoangiogenesis (pathologic generation of the new blood vessels) and extracellular matrix expansion have been described. The vascular endothelial growth factor A (VEGF) has been linked to angiogenesis, but the role of VEGF in DN has not been elucidated yet. VEGF signals mainly through VEGF receptor 2 (VEGFR2). VEGFR2 interacts with alphaV beta3 integrin (AVB3) in kidney. Additionally tenascin C is expressed in the extracellular matrix. Tenascin C and the tenascin C/AVB3 complex have also been linked to angiogenesis, however their roles have not been unveiled yet in the DN. Investigators hypothesize that VEGF signaling and tenascin C play an important role in DN and that VEGFR2, AVB3 and tenascin C interact. The purposes of this study is to characterize social, environmental and biological factors implicated in the DN in Ecuador and define the role of VEGF signaling and tenascin C in the pathogenesis of the DN. Investigators propose to study factors involved in DN in diabetic and non-diabetic adults from general population, with and without DN. In a single time investigators will evaluate demographics data, habits, personal and family history through a survey. Investigators will measure anthropometrics parameters and blood pressure; investigators will quantify blood glucose, glycosylated hemoglobin A1c and proteinuria. In addition investigators will examine the role of tenascin C and VEGF signaling by analyzing paraffin embedded kidney tissue, plasma and urine samples. Characterizing the factors involved in the DN from Hispanic people is key to establish adequate strategies of prevention, diagnosis and treatment in this population. Furthermore elucidating the role of proteins involved in DN may offer valuable tools for the development of new treatments.

DETAILED DESCRIPTION:
1. Determinations of social, environmental and biological factor implicated in diabetic nephropathy in Ecuador Investigators will study subjects from the general population. Investigators will contact community and religious leaders in order to invite adult subjects from the general population to participate in this study and 10000 persons will be enrolled.

   After teaching basic concepts about prevention of diabetic nephropathy in all subjects, investigators will collect demographics data, house conditions and localization (rural, urban or around the cities), number of people that share a home, education level, employment and economical condition, personal health insurance, medical checkup history, toxic habits (alcohol, cigarette abuse of addictive substances) and physical exercises habits. Investigators will collect personal and family antecedent of diabetes mellitus, diabetic nephropathy, hypertension, kidney diseases, diabetes gestational, current treatments and other chronic diseases. Investigators will measure body weight (Kg), height (m) and investigators will calculate body mass index. Investigators will also measure blood pressure, blood glucose, glycosylated hemoglobin, microalbuminuria and proteinuria. Trained personnel will fill out the person's survey. Investigators will supervise and collect data from 2% of the sample.
2. Role of extracellular matrix proteins and growth factors signaling in diabetic nephropathy

   1. Systemic and urine studies: proteins involved in diabetic nephropathy pathogenesis as vascular endothelial factor A (VEGF) and extracellular matrix protein as tenascin C (tenascin) concentration will be measured by a commercially available kits in plasma and urine (respectively). Samples will be obtained from diabetics with (n: 20) and without diabetic nephropathy (n: 20) and from non-diabetic subjects (controls) from the general population (n: 2000). Determinations of social, environmental and biological factor will be completed as in aim 1.
   2. Kidney tissue studies: investigators will determine the role of protein involved in diabetic nephropathy, VEGF signaling and tenascin in:

I) Paraffin embedded kidney tissue obtained from the sample libraries of pathology laboratories will be studied. Slides from non-diabetics (n: 10) and diabetics with diabetic nephropathy (n: 20) and without diabetic nephropathy (n: 10) will be collected. The role of proteins involved in diabetic nephropathy as VEGF signaling and tenascin will be studied by immunohistochemistry and proximity link assay.

II) Paraffin embedded kidney slides from diabetics with diabetic nephropathy (n: 12), non-diabetic control (n: 6) with primary glomerulopathy as minimal change disease, and diabetic controls without diabetic nephropathy (n: 6), will be studied. Investigators will recruit patients with kidney biopsy indicated, and scheduled to be performed, by their medical doctors. After pathology diagnosis completion, some of the remnant paraffin embedded tissue will be used for this study. The role of proteins involved in diabetic nephropathy, VEGF signaling and tenascin will be studied by immunohistochemistry and proximity link assay. Urine and plasma will be collected prior to the kidney biopsy in order to measure protein concentration of potentially useful biomarkers of diabetic nephropathy; VEGF and tenascin levels will be quantified. Patients will be informed and signed consent will be required.

Blood glucose will be measured by the blood glucose meter and test strip. Glycosylated hemoglobin A1c and microalbuminuria (albumin/creatinine in spot urine) will be quantified using the portable machine (Siemens).

In fasting conditions investigators will consider normal blood glucose values <99 mg%, pre-diabetes between 100 and 125 mg% and diabetes ≥126 mg%. In non-fasting conditions values of blood glucose >200mg% will be considered as diabetes. Investigators will deem normal glycosylated A1c hemoglobin values <5.6 %, pre-diabetes between 5.7 and 6.4% and diabetes ≥6.5%.

Investigators will deem normal albuminuria values of albumin/creatinine ratio <29mg/g, microalbuminuria values between 30 and 299 mg/g and macro-albuminuria values ≥300mg/g. Proteinuria will also be evaluated by reactive urine strips.

In the case of inconsistent results or out of range values the analysis will be repeated in the same sample or re analyzed by standard laboratory equipment and techniques.

Investigators will consider diabetic nephropathy as persistent proteinuria associated to diabetic retinopathy and decreased endogen glomerular filtration rate (in subjects without a diagnosis of other kidney or urinary tract diseases). In Type 1 diabetics, diabetic nephropathy will be diagnosed if the history of diabetes is longer than 10 years prior to the onset of proteinuria; in diabetic type 2, proteinuria associated to a decreased glomerular filtration rate at diagnosis time, investigators will deem diabetic nephropathy.

In all paraffin embedded kidney samples we will measure the protein expression and localization. Investigators will use kits, primary and secondary antibodies commercially available to perform immunohistochemistry and proximity link assay. Investigators will perform those experiments in cooperation with pathologist.

All subjects recruited from general population will be identified by a unique code. Number and capital letters code will be placed in the survey and in the sample labels as M0001 (M: city, number 0001: person number 0001). Data will be uploaded and saved in a secure data base. Trained personnel will be in charge of handling the data base. Investigators will supervise the data entry. An investigator at least once every 6 months will randomly select 2% survey and will match it against the information uploaded in the database. Furthermore, investigators will analyze and report all collected data from the surveys even if they are incomplete by adjusting the analysis parameters of the incomplete ones.

Investigators will use descriptive statistic tools to describe groups (mean, standard deviation and standard error or median and interquartile range). For group comparisons, unpaired T test, Mann Whitney or Fisher's test will be used. ANOVA, Kruskal Wallis and Chi Square test will be performed for to compare unmatched groups; to quantify association between two variables Pearson and Spearman correlation test will be used. Simple or multiple regressions will be considered to predict value from variables. P value <0.05 will be deemed significant. A sample from the general population was calculated considering the adult population between 21-70 years old in Ecuador.

ELIGIBILITY:
Inclusion Criteria:

* adults,
* age between 21 and 70 years old,
* persons able to sign informed consent,
* diabetics without diabetic nephropathy,
* diabetic with diabetic nephropathy,
* not hospitalized,
* not suffering acute disease,
* living in their home for at least 6 months before to be contacted.

Exclusion Criteria:

* subjects with acute diseases,
* subjects with not metabolic compensation,
* persons temporarily residing in the place of contact,
* younger than 21 years old,
* older than 70 years old.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample (general healthy population and diabetics subjects), and patients with and without diabetic nephropathy evaluated at Hospital Luis Vernaza
Sampling Method: Non-Probability Sample
Enrollment: 10064 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
House localization | up to 12 month
  House localization (rural, urban or around the cities) in 2000 persons

SECONDARY OUTCOMES:
Protein expression | up to 24 month
  Protein expression in 1000 persons

OTHER OUTCOMES:
Education level | up 12 month
  Education level (primary school, secondary school, university) in 2000 persons.
Employment | up to 12 month
  Employment conditions in 2000 persons.
Health insurance coverage | 12 month
  Personal health insurance coverage in 2000 persons.
Smoking habit | up to 12 month
  Smoking habit in 2000 persons.
Physical exercises habits. | upt to 12 month
  Physical exercises habits in 2000 persons.
Personal and family antecedent of diabetes mellitus | up to 12 month
  Personal and family antecedent of diabetes mellitus in 2000 persons
Personal and family antecedent of kidney diseases | up to 12 month
  Personal and family antecedent of kidney diseases in 2000 persons
Body mass index | up to 12 month
  Body mass index evaluation in 2000 persons
Systolic pressure | 12 month
  Systolic pressure evaluation in 2000 persons
Blood glucose | up 12 month
  Blood glucose evaluation in 2000 persons
Albuminuria | up to 12 month
  Albuminuria evaluation in 2000 persons

CONTACTS AND LOCATIONS:
Overall Officials: Delma Veron, MD PhD, Principal Investigator — Universidad Estatal de Milagro
Locations (1):
- UNEMI, Universidad Estatal de Milagro, Facultad de Ciencias de la Salud, Milagro, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided